CLINICAL TRIAL: NCT05457348
Title: Effect of Single Incision Versus Three Planned Incision to Reduce Pre-operative Astigmatism After Phacoemulsification.
Brief Title: Effect of Single Incision Versus Three Planned Incisions to Reduce Pre-operative Astigmatism After Phacoemulsification.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suleman Roshan Medical College (Other)
Responsible Party: Principal Investigator, Jamshad Ahmed, Professor, Suleman Roshan Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Corneal incision & Astigmatism
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Astigmatism of Both Eyes
Keywords: Astigmatism. phacoemulsification, corneal incision

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into experimental and controlled groups
Who Masked: Participant
Masking Description: The patient will be selected and randomized into two groups after obtaining informed consent. patient will not know about the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A:experimental group (Experimental): those who receive planned incisions
  Interventions: Procedure: Planned incisions during phacoemulsification
- Group B:Controlled group (Active Comparator): the patients who were operated by conventional phacoemulsification
  Interventions: Procedure: Planned incisions during phacoemulsification

INTERVENTIONS:
Procedure: Planned incisions during phacoemulsification — Planned three (one 2.8 mm and two 2.0mm) on the or near to steep meridian will be performed in the experimental group during phacoemulsification

SUMMARY:
Cataract surgery by phacoemulsification is the most commonly performed procedure in Pakistan. Cataract surgery aims for visual rehabilitation and freedom from all kinds of eyewear. Pre-operative corneal astigmatism greater than 1.0 Diopter is reported in 42% preoperatively and 58%postoperatively after implanting a monofocal intraocular lens(IOL). Visual acuity tended to worsen postoperatively with increased astigmatism4. Different treatment modalities are used to reduce astigmatism, like toric IOL. Limbal relaxing incision, actuate keratotomy, intrastromal rings, Lasik and femtosecond laser. Most of these modalities are expensive, so they cannot be afforded by the patients as Pakistan is a low-income country with a per capita income of US$1,562 (160th worldwide)

DETAILED DESCRIPTION:
According to the 2020 estimate, 33·6 million adults aged 50 years and older were blind with cataracts as a leading cause (15·2 million cases). According to Pakistan national blindness survey, cataract is the leading cause of blindness in Pakistan. Cataract surgery by phacoemulsification is the most commonly performed procedure in Pakistan. Cataract surgery aims for visual rehabilitation and freedom from all kinds of eyewear. Pre-operative corneal astigmatism greater than 1.0 Diopter is reported in 42% preoperatively and 58%postoperatively after implanting a mono-focal intraocular lens(IOL). Visual acuity tended to worsen postoperatively with increased astigmatism. Different treatment modalities are used to reduce astigmatism, like toric IOL. Limbal relaxing incision, actuate keratotomy, intrastromal rings, Lasik and femtosecond laser. Most of these modalities are expensive, so they cannot be afforded by the patients as Pakistan is a low-income country with a per capita income of US$1,562 (160th worldwide). Our study aims to compare the results of phacoemulsification cataract surgery with a planned three (one 2.8 mm and two 2.0mm) on the or near to steep meridian incisions ( group A) with convention supero-temporal 2.8 mm clear corneal incision(Group B) for the correction of postoperative astigmatism. We hypothesize that a planned three (one 2.8 mm and two 2.0mm) on the or near to steep meridian incisions ( group A) is better than conventional supero-temporal 2.8 mm clear corneal incision(Group B) for the correction of postoperative astigmatism at a significant level of 0.05.

ELIGIBILITY:
Inclusion Criteria: Cataract patients aged between 50 and 80 years having 1.0 diopters (D) or greater of regular corneal astigmatism documented by keratometry.

Exclusion Criteria:

1. Previous ocular surgery. 2. previous ocular trauma. 3. Pre-existing ocular disease. 4. High intraocular pressure (IOP) 5. Corneal opacity. 6. Strabismus 7. Amblyopia 8. Diabetes mellitus 9. Irregular astigmatism.

-

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-07-30 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-03-02 (Estimated)

PRIMARY OUTCOMES:
Reduction in Astigmatism | Patients will be assessed at first postoperative day then after one month , three months and six months.
  Postoperative reduction in astigmatism after phacoemulsification.

CONTACTS AND LOCATIONS:
Overall Officials: Jamshad Ahmed, FCPS, Principal Investigator — Suleman Roshan Medical College
Locations (1):
- Suleman Roshan Medical College Hospital, Tando Adam, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
the clinical study report will be shared with all participants if they desire. the study will be published in a journal. it will be available to all participants and the research community.
Supporting Information: CSR
Time Frame: after 6 months
Access Criteria: contact with principal investigator

REFERENCES:
- [Result] GBD 2019 Blindness and Vision Impairment Collaborators; Vision Loss Expert Group of the Global Burden of Disease Study. Causes of blindness and vision impairment in 2020 and trends over 30 years, and prevalence of avoidable blindness in relation to VISION 2020: the Right to Sight: an analysis for the Global Burden of Disease Study. Lancet Glob Health. 2021 Feb;9(2):e144-e160. doi: 10.1016/S2214-109X(20)30489-7. Epub 2020 Dec 1. PMID 33275949
- [Result] Dineen B, Bourne RR, Jadoon Z, Shah SP, Khan MA, Foster A, Gilbert CE, Khan MD; Pakistan National Eye Survey Study Group. Causes of blindness and visual impairment in Pakistan. The Pakistan national blindness and visual impairment survey. Br J Ophthalmol. 2007 Aug;91(8):1005-10. doi: 10.1136/bjo.2006.108035. Epub 2007 Jan 17. PMID 17229806
- [Result] Liu YC, Wilkins M, Kim T, Malyugin B, Mehta JS. Cataracts. Lancet. 2017 Aug 5;390(10094):600-612. doi: 10.1016/S0140-6736(17)30544-5. Epub 2017 Feb 25. PMID 28242111
- [Result] Day AC, Dhariwal M, Keith MS, Ender F, Perez Vives C, Miglio C, Zou L, Anderson DF. Distribution of preoperative and postoperative astigmatism in a large population of patients undergoing cataract surgery in the UK. Br J Ophthalmol. 2019 Jul;103(7):993-1000. doi: 10.1136/bjophthalmol-2018-312025. Epub 2018 Sep 6. PMID 30190365
- [Result] Ren Y, Fang X, Fang A, Wang L, Jhanji V, Gong X. Phacoemulsification With 3.0 and 2.0 mm Opposite Clear Corneal Incisions for Correction of Corneal Astigmatism. Cornea. 2019 Sep;38(9):1105-1110. doi: 10.1097/ICO.0000000000001915. PMID 30844842
- [Result] What is current GDP of Pakistan?. Paid for articles.com. naeemofficial3; Jun 19, 2022
- See also: link for first reference — https://doi.org/10.1016/s2214-109x(20)30489-7
- See also: link for second reference — https://doi.org/10.1136/bjo.2006.108035
- See also: link for third reference — https://doi.org/10.1016/s0140-6736(17)30544-5
- See also: link for fifth reference — https://doi.org/10.1097/ico.0000000000001915